CLINICAL TRIAL: NCT03565731
Title: A Novel Behavioral Approach for the Adoption and Maintenance of Habitual Physical Activity
Brief Title: Exercise Values of Life and Vitality Everyday
Acronym: EVOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2059-17; 1R03DK114254 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2018-06-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Physical Activity; Lifestyle; Behavior; Lifestyle, Sedentary; Acceptance and Commitment Therapy; Exercise; ACT
MeSH Terms: conditions — Motor Activity; Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-PA Intervention (Experimental): The primary goal of the intervention is to increase values-based autonomous motivation to increase bout-related MVPA using a single workshop. Participants will engage in basic and advanced values clarification exercise to help clarify (1) the relative importance of major values domains (e.g. social, vocational, recreational), and (2) the potential role of PA in empowering functioning in these domains. Participants will generate their own activity goals and additional values-based goals. In addition, acceptance strategies will be taught to reduce cognitive and emotional barriers to meeting values-based goals. Participants will be asked to report progress on goals each week via an automated email survey from a secure project website. Upon completing the survey, participants will receive standardized responses via email. Monthly phone calls will be brief, semi-structured, and designed to review key principles and trouble-shoot specific barriers identified by the participant.
  Interventions: Behavioral: ACT-PA

INTERVENTIONS:
Behavioral: ACT-PA — The overall goal of the intervention is to increase bout-related moderate-to-vigorous physical (MVPA) activity to greater than 200 minutes per week. The basic structure is an initial on-site, group-based intervention workshop, written materials, weekly emails, and monthly phone calls for a total of 3 months.

SUMMARY:
The purpose of this study is to develop and test a brief program to help overweight people become more physically active. We plan to design a program that teaches people how to become more active by identifying how fitness enables them to live their lives better.

Participants will be asked to complete questionnaires and wear a device that tracks their exercise for 1 week. If accepted into the study, they will receive a 1 day program designed to help them exercise more. Then they will receive phone calls and emails for support after the program. Finally, participants will come in 3 and 6 months after the program to complete the same questionnaires and wear the exercise tracker again.

The study is primarily interested in increasing exercise levels, and so we hope to see participants exercising more after the program than they were before. We will also ask them questions (via the questionnaires) that tell us the degree to which they are exercising based on their one desires and values, as opposed to doing it because they were told to.

DETAILED DESCRIPTION:
Despite the importance of adoption and maintenance of habitual moderate to vigorous-intensity physical activity (MVPA) for health benefits and long-term weight management, current comprehensive lifestyle interventions place little emphasis on physical activity behavior change strategies and have only modest impact on MVPA. Acceptance and Commitment Therapy (ACT), a well validated, newer generation behavioral approach uses values of clarification and commitment strategies, along with acceptance-based skills training, to effect health behavior change that is consistent with personally identified values. ACT presents a theoretically consistent and potentially powerful intervention framework from which to target values-based autonomous motivation and increase MVPA. The overall aim of this study is to test the feasibility, acceptability, and preliminary efficacy of an ACT-based workshop intervention for increasing bout-related MVPA for overweight and obese, insufficiently active adults using a single-arm design. We will recruit 48 overweight/obese, insufficiently active adults across multiple cohorts and provide them with a 4-hour, ACT-based workshop followed by weekly emails and monthly phone calls for 3 months. The primary goal of the workshop is to use values clarification and acceptance-based skills training to increase values-based autonomous motivation and bout-related MVPA. Participants will self-monitor and report on progress via weekly emails and monthly phone calls. Assessments will be at baseline, 3, and 6 months. The goal of this study is threefold: 1) to determine the feasibility and acceptability of the ACT workshop intervention by assessing the completion of the intervention at all time points and via questionnaires; 2) to show changes in autonomous motivation and values-consistent behavior at the end of the intervention; and 3) to show changes in physical activity, by use of an objectively measured physical activity devices, where participants are engaging in at least 200 minutes of MVPA at 3 and 6-months)

This study will be conducted at the Miriam Hospital Weight Control and Diabetes Research Center by Drs. Jason Lillis and Dale Bond.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25-45 kg/m2
* Report being insufficiently active (i.e., <150 minutes per week of bout related MVPA)

Exclusion Criteria:

* Unable to engage in physical activity safely due to medical status
* Unable to read or understand study materials
* Currently in another physical activity or weight control program
* Currently taking medications that cause dizziness or feeling faint while standing (e.g., some hypertension medications
* Report any condition that would preclude adherence to the intervention protocol (e.g., current or past substance use disorder or psychiatric hospitalization)
* Plans to relocate during the study timeline
* Terminal illness diagnosis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change in bout-related moderate to vigorous physical activity (MVPA) | Change from baseline to 3 and 6 months
  Average daily minutes spent in objectively measured, bout-related MVPA assessed via a multi-sensor activity monitoring device.

SECONDARY OUTCOMES:
Feasibility of the ACT workshop intervention | End of 3-month intervention
  Successful completion of ≥70% of email surveys and intervention phone calls
Acceptability of the ACT workshop intervention | End of 3-month intervention
  An adapted, 15-item version of a previous validated feasibility and acceptability measure for PA interventions with a five-point Likert scale (1 = "don't agree at all" to 5 = "totally agree"). Item examples will include, "I enjoyed participating in the intervention," "I think the intervention strategies were appropriate," and, "I found the lessons to be easy to understand."
Change in autonomous motivation | Change from baseline to 3 and 6 months
  Exercise Self-Regulation Questionnaire. A 12-item, Likert scaled ("not true at all" to "very true") measure that assesses why a respondent engages in PA by providing several possible reasons that represent varying degrees of autonomous motivation.
Change in values-consistent behavior | Change from baseline to 3 and 6 months
  Comprehensive Assessment of Acceptance and Commitment Therapy Processes Questionnaire. A 23-item measure with a values subscale that assesses whether individuals are living consistent with their values and what barriers are getting in the way

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Lillis J, Bond DS. Values-based and acceptance-based intervention to promote adoption and maintenance of habitual physical activity among inactive adults with overweight/obesity: a study protocol for an open trial. BMJ Open. 2019 Jan 9;9(1):e025115. doi: 10.1136/bmjopen-2018-025115. PMID 30782749